CLINICAL TRIAL: NCT05474469
Title: Effects of Diaphragmatic Breathing With and Without Abdominal Muscles Strength Training Program on Pelvic Floor Strength, Endurance and Quality of Life in Postnatal Women
Brief Title: Diaphragmatic Breathing With and Without Abdominal Muscles Strength Training Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0509
Record Dates: First submitted 2022-07-24; First posted 2022-07-26 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Pelvic Floor Muscle Weakness; Endurance; Quality of Life
Keywords: Abdominal Muscles; Breathing Exercises; Exercise; Pelvic Floor; Quality Of Life
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diaphragmatic breathing in combination with abdominal muscle strengthening exercises (Experimental): Exprimental Group ( Group A) will receive diaphragmatic breathing in combination with abdominal muscle strengthening exercises .12 treatment sessions for 4 weeks period, which consisted of 03 treatment sessions per week.
  Interventions: Other: Diaphragmatic breathing exercises; Other: Abdominal muscle strengthening exercises
- Diaphragmatic breathing Exercises only without abdominal muscle strengthening exercises (Active Comparator): Active comparator (Group B) will receive diaphragmatic breathing only. 12 treatment sessions for 4 weeks period, which consisted of 03 treatment sessions per week.
  Interventions: Other: Diaphragmatic breathing exercises

INTERVENTIONS:
Other: Diaphragmatic breathing exercises — 12 treatment sessions for 4 weeks period, which consisted of 03 treatment sessions per week.
Other: Abdominal muscle strengthening exercises — 12 treatment sessions for 4 weeks period, which consisted of 03 treatment sessions per week.
  Arms: Diaphragmatic breathing in combination with abdominal muscle strengthening exercises

SUMMARY:
The postpartum period is excessively weak and have hypotonic abdominal muscles, making the ligaments and connective tissue softer and more elastic. The importance of exercise in the postpartum period is very important in this regard.

This study will be a Randomized control trial used to compare the effects of diaphragmatic breathing with and without abdominal muscles strength training program on pelvic floor strength and endurance and quality of life in postnatal women. Subjects meeting the inclusion and exclusion criteria will be divided into two groups using lottery method. Assessment will be done using PERFECT scheme questionnaire and SF- 36 quality of life questionnaire. Subjects in one group will receive diaphragmatic breathing exercises along with pelvic muscle strength training and subjects in other group will receive only diaphragmatic breathing exercises. Each subject will receive 12 treatment sessions for 4 weeks. Results will be analyzed for any change by using SPSS25.

DETAILED DESCRIPTION:
The postpartum period is excessively weak and have hypotonic abdominal muscles, making the ligaments and connective tissue softer and more elastic. These changes result in anatomical, physiological and biomechanical alterations. Therefore, these factors are responsible for the lack of necessary support for the waist region, pain, disability and negative impact on health-related quality of life. The importance of exercise in the postpartum period is very important in this regard. Postnatal exercises have several benefits such as improving pelvic floor strength and endurance and quality of life and increasing the general well-being, preventing the diastasis of the rectus Abdominis muscle (RAM) increasing cardiovascular endurance and bone mineral density.

This study will be a Randomized control trial used to compare the effects of diaphragmatic breathing with and without abdominal muscles strength training program on pelvic floor strength and endurance and quality of life in postnatal women. Subjects meeting the inclusion and exclusion criteria will be divided into two groups using lottery method. Assessment will be done using PERFECT scheme questionnaire and SF- 36 quality of life questionnaire. Subjects in one group will receive diaphragmatic breathing exercises along with pelvic muscle strength training and subjects in other group will receive only diaphragmatic breathing exercises. Each subject will receive 12 treatment sessions for 4 weeks. Results will be analyzed for any change by using SPSS25.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 35 years.
* Women between 2 to 6 months post-natal.
* Women with stable somatic state.
* Women with no cognitive dysfunction.

Exclusion Criteria:

* Women with respiratory problems.
* Women with severe back pain.
* Patients with any pelvic pathology
* Patient with any previous neurological disorders

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Postnatal Women
Enrollment: 74 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
PERFECT scheme questionnaire | 4 Weeks
  The term PERFECT stands for power (or pressure), endurance (E), repetitions (R), rapid contractions (F), and lastly, every contraction timed (ECT). The Pelvic Floor Muscle Assessment Scheme was created to streamline and explain the process. This program may provide suggestions for developing patient-specific exercise plans that correspond to the principles of muscle training."
SF-36 quality of life questionnaire | 4 Weeks
  Physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH) are the eight scales that the SF-36 measures. Different amounts from each scale do go into the scoring of the PCS and MCS measures.

CONTACTS AND LOCATIONS:
Overall Officials: Sabiha Arshad, M.Phil, Principal Investigator — Riphah International University
Locations (1):
- Islamic Center Sialkot, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gursen C, Inanoglu D, Kaya S, Akbayrak T, Baltaci G. Effects of exercise and Kinesio taping on abdominal recovery in women with cesarean section: a pilot randomized controlled trial. Arch Gynecol Obstet. 2016 Mar;293(3):557-65. doi: 10.1007/s00404-015-3862-3. Epub 2015 Sep 2. PMID 26329802
- [Background] Ashton-Miller JA, DeLancey JO. Functional anatomy of the female pelvic floor. Ann N Y Acad Sci. 2007 Apr;1101:266-96. doi: 10.1196/annals.1389.034. Epub 2007 Apr 7. PMID 17416924
- [Background] Bernardes BT, Resende AP, Stupp L, Oliveira E, Castro RA, Bella ZI, Girao MJ, Sartori MG. Efficacy of pelvic floor muscle training and hypopressive exercises for treating pelvic organ prolapse in women: randomized controlled trial. Sao Paulo Med J. 2012;130(1):5-9. doi: 10.1590/s1516-31802012000100002. PMID 22344353
- [Background] Janakiraman B, Gebreyesus T, Yihunie M, Genet MG. Knowledge, attitude, and practice of antenatal exercises among pregnant women in Ethiopia: A cross-sectional study. PLoS One. 2021 Feb 19;16(2):e0247533. doi: 10.1371/journal.pone.0247533. eCollection 2021. PMID 33606844
- [Background] Oliveira MC, Oliveira M, Silva H, Gomes A, Nascimento G, Marini G, Micussi MT. Evaluation of satisfaction of pelvic floor muscle training isolated and associated with tibial nerve stimulation in women with mixed urinary incontinence: A randomized, single-blinded clinical trial. Eur J Obstet Gynecol Reprod Biol. 2021 Oct;265:60-65. doi: 10.1016/j.ejogrb.2021.06.024. Epub 2021 Jun 24. PMID 34461383